CLINICAL TRIAL: NCT04340141
Title: A Phase III Trial of Perioperative Versus Adjuvant Chemotherapy for Resectable Pancreatic Cancer
Brief Title: Testing the Use of the Usual Chemotherapy Before and After Surgery for Removable Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A021806; NCI-2020-01560 (Registry Identifier: NCI Clinical Trial Reporting Program); U10CA180821 (NIH)
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Adenosquamous Carcinoma; Resectable Pancreatic Adenocarcinoma; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (perioperative chemotherapy, surgery) (Experimental): Patients receive oxaliplatin intravenously (IV) over 2 hours, irinotecan hydrochloride IV over 90 minutes, and leucovorin calcium over 2 hours on day 1, and fluorouracil IV over 46-48 hours on days 1-3. Treatment repeats every 14 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Within 2-8 weeks of completing neoadjuvant chemotherapy, patients undergo surgical resection. Patients then receive oxaliplatin IV over 2 hours, irinotecan hydrochloride IV over 90 minutes, and leucovorin calcium over 2 hours on day 1, and fluorouracil IV over 46-48 hours on days 1-3. Treatment repeats every 14 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan Hydrochloride; Drug: Leucovorin Calcium; Drug: Fluorouracil; Procedure: Resection; Other: Questionnaire Administration
- Arm II (surgery, adjuvant chemotherapy) (Active Comparator): Patients undergo surgical resection. Beginning 3-12 weeks after surgery, patients then receive oxaliplatin IV over 2 hours, irinotecan hydrochloride IV over 90 minutes, and leucovorin calcium over 2 hours on day 1, and fluorouracil IV over 46-48 hours on days 1-3. Treatment repeats every 14 days for 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan Hydrochloride; Drug: Leucovorin Calcium; Drug: Fluorouracil; Procedure: Resection; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Oxaliplatin — Given IV
Drug: Irinotecan Hydrochloride — Given IV
Drug: Leucovorin Calcium — Given IV
Drug: Fluorouracil — Given IV
Procedure: Resection — Undergo surgical resection
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial compares perioperative chemotherapy (given before and after surgery) versus adjuvant chemotherapy (given after surgery) for the treatment of pancreatic cancer that can be removed by surgery (removable/resectable). Chemotherapy drugs, such as fluorouracil, irinotecan, leucovorin, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy before and after surgery (perioperatively) may work better in treating patients with pancreatic cancer compared to giving chemotherapy after surgery (adjuvantly).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate and compare overall survival (OS) in patients with resectable pancreatic adenocarcinoma treated with perioperative fluorouracil, irinotecan hydrochloride, leucovorin calcium and oxaliplatin (modified [m]FOLFIRINOX) and surgery versus up-front surgery followed by adjuvant mFOLFIRINOX.

SECONDARY OBJECTIVES:

I. To evaluate and compare disease-free survival (DFS) in patients with resectable pancreatic adenocarcinoma treated with perioperative mFOLFIRINOX and surgery versus up-front surgery followed by adjuvant mFOLFIRINOX.

II. To evaluate and compare time to locoregional recurrence (TLR) in patients with resectable pancreatic adenocarcinoma treated with perioperative mFOLFIRINOX and surgery versus up-front surgery followed by adjuvant mFOLFIRINOX.

III. To evaluate and compare time to distant metastases (TDM) in patients with resectable pancreatic adenocarcinoma treated with perioperative mFOLFIRINOX and surgery versus up-front surgery followed by adjuvant mFOLFIRINOX.

IV. To evaluate and compare the R0 resection rate in patients with resectable pancreatic adenocarcinoma treated with perioperative mFOLFIRINOX and surgery versus up-front surgery followed by adjuvant mFOLFIRINOX.

V. To evaluate and compare rate of unresectability in patients with resectable pancreatic adenocarcinoma treated with perioperative mFOLFIRINOX and surgery versus up-front surgery followed by adjuvant mFOLFIRINOX.

VI. To evaluate rate of pathologic complete response in patients randomized to the perioperative therapy arm.

VII. To evaluate and compare mFOLFIRINOX dose intensity delivered and number of cycles received in patients with resectable pancreatic adenocarcinoma treated with perioperative mFOLFIRINOX and surgery versus up-front surgery followed by adjuvant mFOLFIRINOX.

VIII. To evaluate and compare adverse event profile in patients with resectable pancreatic adenocarcinoma treated with perioperative mFOLFIRINOX and surgery versus up-front surgery followed by adjuvant mFOLFIRINOX.

IX. To compare physical functioning, nausea/vomiting, and diarrhea, as measured with the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) between patients with resectable pancreatic adenocarcinoma treated with perioperative mFOLFIRINOX and surgery versus up-front surgery followed by adjuvant mFOLFIRINOX.

X. To prospectively assess the influence of diet, body mass index, weight loss, physical activity, and other lifestyle habits on the disease-free survival and overall survival among patients with localized pancreatic cancers.

XI. To assess the influence of diet, obesity, physical activity, and other lifestyle habits on the risk of toxicity associated with chemotherapy.

XII. To evaluate the ability of computed tomography (CT)-based radiomics in distinguishing post-neoadjuvant chemotherapy (NAC) fibrosis from viable tumor in patients randomized to the perioperative therapy arm.

XIII. To determine whether CT-based radiomics retrieved from baseline examination may act as non-invasive predictors of survival outcome in patients randomized to the adjuvant therapy arm.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive oxaliplatin intravenously (IV) over 2 hours, irinotecan hydrochloride IV over 90 minutes, and leucovorin calcium over 2 hours on day 1, and fluorouracil IV over 46-48 hours on days 1-3. Treatment repeats every 14 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Within 2-8 weeks of completing neoadjuvant chemotherapy, patients undergo surgical resection. Patients then receive oxaliplatin IV over 2 hours, irinotecan hydrochloride IV over 90 minutes, and leucovorin calcium over 2 hours on day 1, and fluorouracil IV over 46-48 hours on days 1-3. Treatment repeats every 14 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Patients undergo surgical resection. Beginning 3-12 weeks after surgery, patients then receive oxaliplatin IV over 2 hours, irinotecan hydrochloride IV over 90 minutes, and leucovorin calcium over 2 hours on day 1, and fluorouracil IV over 46-48 hours on days 1-3. Treatment repeats every 14 days for 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 6 years.

ELIGIBILITY:
Inclusion Criteria:

PRE-REGISTRATION:

* Pathology: Histologic or cytologic proof of pancreatic adenocarcinoma or adenosquamous carcinoma
* TNM Stage: Tx-4, N0-1, M0 (M0 disease does not include spread to distant lymph nodes and organs)
* Resectable Primary Tumor: Local radiographic reading must be consistent with resectable disease defined as the following on 1) arterial and venous phase contrast-enhanced abdominal/pelvic CT scan or abdominal/pelvic magnetic resonance imaging (MRI) scan and 2) chest CT:

  * No involvement or abutment of the celiac artery, common hepatic artery, superior mesenteric artery, or replaced right hepatic artery (if applicable)
  * Less than 180 degree interface between tumor and vessel wall of the portal vein or superior mesenteric vein, and patent portal vein/splenic vein confluence
  * No evidence of metastatic disease
* Measurable disease or non-measurable disease o Non-measurable disease is defined as cytologic or histologic confirmation of adenocarcinoma of adenosquamous carcinoma by fine needle aspiration or core-biopsy of the pancreas without measurable disease by radiographic imaging

REGISTRATION:

* Confirmation of resectable disease by real-time central imaging review by the Alliance Imaging Core Lab at Imaging and Radiation Oncology Core (IROC) Ohio
* Determined to be appropriate candidate for curative-intent pancreatectomy by surgeon intending to perform the resection
* No prior radiation therapy, chemotherapy, targeted therapy, investigational therapy, or surgery for pancreatic cancer
* Not pregnant and not nursing, because this study involves an agent that has known genotoxic, mutagenic, and teratogenic effects.
* Therefore, for women of childbearing potential only, a negative pregnancy test done =< 14 days prior to registration is required
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Total Neuropathy Score < 2
* Absolute neutrophil count (ANC) >= 1,500/uL
* Platelet count >= 100,000/uL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (If obstructive jaundice is present, then biliary drainage must be initiated and total bilirubin =< 3.0)
* Creatinine =< 1.5 x ULN OR calculated (Calc.) creatinine clearance >= 30 mL/min (Calculated using the Cockcroft-Gault equation)
* No known Gilbert's Syndrome or known homozygosity for UGAT1A1*28 polymorphism
* No comorbid conditions that would prohibit curative-intent pancreatectomy
* Chronic concomitant treatment with strong inhibitors of CYP3A4 is not allowed on this study. Patients on strong CYP3A4 inhibitors must discontinue the drug prior to registration
* Chronic concomitant treatment with strong inducers of CYP3A4 is not allowed on this study. Patients on strong CYP3A4 inducers must discontinue the drug prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Time between randomization and death from any cause, assessed up to 6 years.
  Overall survival is defined as the time from randomization to death due to any cause. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator. The treatment arms will be compared using a stratified Cox regression model, and hazard ratios from each arm will be estimated.

SECONDARY OUTCOMES:
Disease-free survival (DFS) | Time between randomization and progression prior to surgery, metastases detected during surgery, recurrence (locoregional and/or distant) after resection, and death due to all causes, assessed up to 6 years.
  Disease-free survival (DFS) is defined as the time from randomization to the date of progression prior to surgery, metastases detected during surgery, recurrence (locoregional and/or distant) after resection, and death due to all causes, whichever occurs first. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time to locoregional recurrence (TLR) | Time between randomization and locoregional recurrence after resection, assessed up to 6 years.
  Time to locoregional recurrence (TLR) is defined as the time from randomization to the date of locoregional recurrence after resection. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time to distant metastases (TDM) | Time between randomization and metastases prior to surgery, metastases detected during surgery, or distant recurrence after resection, assessed up to 6 years.
  Time to distant metastases (TDM) is defined as the time from randomization to the date of metastases prior to surgery, metastases detected during surgery, or distant recurrence after resection. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
R0 resection rate | At time of surgery.
  The rate (percentage) of patients with negative resection margins after undergoing surgery.
Rate of unresectability | At time of surgery or planned time of surgery.
  The rate (percentage) of patients who cannot undergo surgery due to adverse events, progressive disease, death, poor performance, or patient/physician decision, are deemed unresectable before surgery, or resection was not performed during surgery.
Pathologic complete response (pCR) rate | At time of surgery.
  The rate (percentage) of patients who achieve a pathologic complete response (pCR) confirmed by histopathologic review of the surgical specimen.
Incidence of adverse events (AEs), assessed using National Cancer Institute (NCI) common terminology criteria for adverse events (CTCAE) version 5.0 (v5.0) | Up to 2 years.
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine adverse event patterns within treatment arms and during the following three time points: during perioperative chemotherapy, surgical complications during surgery and post-operative period for 30 days, and during adjuvant chemotherapy.
Fluorouracil, irinotecan hydrochloride, leucovorin calcium, and oxaliplatin (modified [m]FOLFIRINOX) dose intensity delivered | 8 months
  Dose intensity is defined as the percentage of total cumulative dose the patient received divided by the total dose planned per protocol times 100.
Fluorouracil, irinotecan hydrochloride, leucovorin calcium and oxaliplatin (modified [m]FOLFIRINOX) number of cycles received | 8 months
  The number of cycles received is defined as the total number of cycles that the participant received at least one dose of any agent in mFOLFIRINOX.
Quality of life as assessed by the physical functioning, nausea/vomiting, and diarrhea subscales in the Quality of Life Questionnaire-Core 30 (QLQ-C30) | 8 weeks
  Quality of Life Questionnaire-Core 30 (QLQ-C30) is a 30-item questionnaire to assess the overall quality of life in cancer patients. QLQ-C30 includes functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting), and other (dyspnoea, appetite loss, insomnia, constipation/diarrhea, and financial difficulties). Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score=better level of physical functioning, greater occurrence of nausea/vomiting, and greater occurrence of diarrhea.
Influence of diet, body mass index, weight loss, physical activity, and other lifestyle habits on overall survival | Time between randomization and death from any cause, assessed up to 6 years.
  Multivariate Cox proportional hazards models will be fit for overall survival (OS) endpoint (defined above) with covariates corresponding to baseline diet and lifestyle questionnaire responses and hazard ratios and 95% confidence intervals will be reported.
Influence of diet, body mass index, weight loss, physical activity, and other lifestyle habits on disease-free survival (DFS) | Time between randomization and progression prior to surgery, metastases detected during surgery, recurrence (locoregional and/or distant) after resection, and death due to all causes, assessed up to 6 years.
  Multivariate Cox proportional hazards models will be fit for disease-free survival (DFS) endpoint (defined above) with covariates corresponding to baseline diet and lifestyle questionnaire responses and hazard ratios and 95% confidence intervals will be reported.
Influence of diet, body mass index, weight loss, physical activity, and other lifestyle habits on the risk of grade 3+ adverse event associated with chemotherapy | Up to 2 years.
  Multivariate Logistic models will be fit for the binary endpoint of grade 3+ adverse event (patient experiences at least one grade 3 or higher adverse event during treatment)
The ability of computed tomography (CT)-based radiomics to distinguish post-neoadjuvant chemotherapy (NAC) fibrosis from viable tumor as measured by comparison to histological evaluation | At time of surgery.
  Comparison between computed tomography (CT)-based radiomics and histological tumor fibrosis proportions will be measured using Spearman's rank correlation coefficient.
Computed tomography (CT)-based radiomics as non-invasive predictors of overall survival | Time between randomization and death from any cause, assessed up to 6 years.
  Multivariate Cox proportional hazards model will be fit for overall survival (OS) endpoint (defined above) with covariates chosen from all available radiomics features using the least absolute shrinkage and selection operator (LASSO) method with 10-fold cross-validation (CV) and additionally adjusted for clinically important confounders. After the final model is selected the area under the receiver operating characteristic curve (AUC) will be reported to indicate the prediction performance of the radiomics model.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina R. Ferrone, MD, Study Chair — Massachusetts General Hospital
Locations (453):
- United States (441):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Thomas Hospital, Fairhope, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Community Cancer Institute, Clovis, California
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Mills Health Center, San Mateo, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - AdventHealth Porter, Denver, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Schulze Family Foundation Cancer Clinic - Bonita Health Center, Bonita Springs, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Tampa General Hospital, Tampa, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Ochsner Hematology Oncology North Shore - Covington (West Region), Covington, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - UM Saint Joseph Medical Center, Towson, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Jersey City Medical Center, Jersey City, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - South Shore University Hospital, Bay Shore, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - The Cancer Institute at Saint Francis Hospital, East Hills, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Northwell Health Cancer Institute at Huntington, Greenlawn, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Upstate Cancer Center at Oswego, Oswego, New York
  - Queens Cancer Center, Rego Park, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - CarolinaEast Medical Center, New Bern, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Avera Cancer Institute - Mitchell, Mitchell, South Dakota
  - Avera Cancer Institute at Pierre, Pierre, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Avera Cancer Institute at Yankton, Yankton, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Inova Loudoun Hospital, Leesburg, Virginia
  - Sentara Leigh Hospital, Norfolk, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (12):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - BCCA-Vancouver Island Cancer Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre/Nova Scotia Health Authority, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes